CLINICAL TRIAL: NCT03125551
Title: Viscoelastic Point-of-Care Coagulation Monitoring and Dietary Supplements: A Randomized, Double-blind, Placebo-controlled Trial
Brief Title: ROTEM and Dietary Supplements
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Study requires Medicines Control council approval
Sponsor: University of Pretoria (Other)
Responsible Party: Principal Investigator, Jayde Wyngaard, Dr, University of Pretoria
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Diagnostic
Other Study IDs: MMed Anaesthesiology -15402364
Record Dates: First submitted 2017-03-27; First posted 2017-04-24 (Actual); Last update posted 2018-05-09 (Actual); Status verified 2018-05

CONDITIONS: Dietary Supplements; Bleeding Tendency; Due to Coagulation Defect
Keywords: Dietary supplements; Bleeding tendency
MeSH Terms: conditions — Hemostatic Disorders | interventions — ginger extract; Ginkgo Extract; Asian ginseng

STUDY DESIGN:
Intervention Model Description: Five- armed, placebo- controlled ( 4 intervention groups and 1 placebo group)
Who Masked: Participant, Outcomes Assessor
Masking Description: Each participant will be blinded to the dietary supplement which they will be taking. The medical technologist doing the ROTEM will be blinded to the dietary supplements as well.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- Ginger (Active Comparator): Ginger ( Zingiber officinale) 4 grams po dly for 14 days
  Interventions: Dietary Supplement: Ginger
- Garlic (Active Comparator): Garlic (Allium sativum) 4-12 mg alliin po dly for 14 days
  Interventions: Dietary Supplement: Garlic
- Ginkgo Biloba (Active Comparator): Ginkgo Biloba 40mg po tds for 14 days
  Interventions: Dietary Supplement: Ginkgo Biloba
- Ginseng (Active Comparator): Ginseng 400mg po dly for 14 days
  Interventions: Dietary Supplement: Ginseng
- Placebo (Placebo Comparator): Placebo po dly for 14 days
  Interventions: Other: Placebo

INTERVENTIONS:
Dietary Supplement: Ginger — Ginger dosage at daily recommended allowance
  Arms: Ginger
Dietary Supplement: Garlic — Garlic dosage at daily recommended allowance
  Arms: Garlic
Dietary Supplement: Ginkgo Biloba — Ginkgo Biloba dosage at daily recommended allowance
  Arms: Ginkgo Biloba
Dietary Supplement: Ginseng — Ginseng dosage at daily recommended allowance
  Arms: Ginseng
Other: Placebo — Daily dosage strategy
  Arms: Placebo

SUMMARY:
Dietary Supplements can affect platelet activation and aggregation, which could result in bleeding tendencies. This study wishes to evaluate the influence that these supplements has on platelet function using Rotational thromboelastometry.

DETAILED DESCRIPTION:
The WHO informs us that more than 80% of patients in Africa use traditional/herbal medicines as their primary source of health care. The Mayo Clinic stated that nearly 40% of adults reported using complementary and alternative medicine (CAM). Many of these herbal medicines as well as dietary supplements have effects on the coagulation cascade and have been identified as such using laboratory tests including aPTT, PT, INR, light transmission aggregometry and impedence aggregometry to mention but a few.

This study wishes to evaluate coagulation abnormalities using viscoelastic point-of-care coagulation monitoring in this population. This test is readily available in large hospitals and academic settings and is increasingly being used in perioperative medicine. It provides information on coagulation and thrombolysis with minimal delay when compared to other laboratory-based coagulation tests.

The dietary supplements which will be evaluated in this study are ginger, garlic, gingko biloba and ginseng. These four herbal supplements were identified as the most commonly used substances known to modulate the coagulation system. These herbal supplements will be investigated within their maximum daily allowance dosages.

A five-armed placebo-controlled study will be undertaken and study subjects will be recruited on a volunteer basis. Subjects will be divided into five groups and each group will receive one of the four dietary supplements and the fifth group placebo, for a two week period. Rotational thromboelastometry (ROTEM) studies will be performed on blood samples obtained from each participant at baseline and at the end of the treatment period to identify coagulation abnormalities. Most of these herbal medicines have been identified to affect platelet function and this study will specifically look at platelet function determined by maximum clot firmness (MCF) in the ROTEM analysis.

Viscoelastic point-of-care coagulation monitoring in patients using herbal medicines and dietary supplements will aid decision making regarding cause of perioperative haemorrhage and need for specific blood products. It will therefore assist with goal-directed management of perioperative haemorrhage. It will also aid the anaesthetist wishing to employ a regional anaesthetic technique in this patient group.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18-60 years
2. Both males and females
3. Healthy volunteers
4. Smokers and Non-smokers
5. Staff frequenting the theatre complex at Steve Biko Academic Hospital

Exclusion Criteria:

1. Use of any medication, excluding oral contraceptive pills, in the two week period prior to commencement of the study. Medicines excluded, include aspirin, dietary supplements, herbal teas, anticoagulants and other non-steroidal anti-inflammatory medications. . Oral contraceptive pills were omitted as an exclusion criteria, taking into account that the majority of woman use these. The results of the study will be a better reflection of the effect of these dietary supplements in the modern day woman. Its coagulant properties will be taken into account during data analysis.
2. History of any chronic medical or psychiatric illness.
3. Current excessive alcohol intake - more than 14 units a week in woman and more than 21 units a week in men.
4. Pregnant or lactating mothers.
5. Possible planned surgery during the study period

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2017-06 (Estimated); Primary Completion 2017-07 (Estimated); Study Completion 2017-08 (Estimated)

PRIMARY OUTCOMES:
Platelet dysfunction determined by ROTEM when consuming ginger, garlic, ginkgo biloba and ginseng. | 2-4 weeks
  To determine if viscoelastic point-of-care coagulation monitoring (ROTEM) detects abnormalities in platelet function when subjects consume ginger, garlic, ginkgo biloba and ginseng within their recommended daily allowances. ExTEM and FibTEM analysis will be performed and difference in MCF values will determine if there is platelet dysfunction or not.

CONTACTS AND LOCATIONS:
Overall Officials: Jayde V Wyngaard, MBCHB, Principal Investigator — University of Pretoria

IPD SHARING:
Plan to Share IPD: No